CLINICAL TRIAL: NCT03787771
Title: The Fecal Microbiota Transplantation Registry
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: FMTR
Record Dates: First submitted 2018-06-27; First posted 2018-12-26 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Fecal Microbiota Transplantation
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FMT recipents: Subject who has received or planning to receive FMT or other gut-related microbiota products in routine clinical practice or research
- FMT donors: Subject who has donated stool or planning to donate stool for FMT or production of other gut-related microbiota products in routine clinical practice or research.

SUMMARY:
The human intestinal microbiota is composed of complex community of 10*13 to 10*14 commensal microorganisms[1]. Human intestine provides a nutrient-rich habitat for intestinal microorganism which allows a diverse ecosystem to enhance their host's immune system and facilitate digestive activities. Numerous researches are investigating the role of gut microbiota in human homeostasis, which may be related to the pathogenesis of gastrointestinal disease and autoimmune disorder.

Fecal microbiota transplantation (FMT) is defined as infusion of feces from healthy donors to affected subjects. FMT works by altering the patient's microbiome and it is now recommended as an effective therapy for Clostridium difficile infection (CDI) not responding to standard therapies[8]. It has attracted great interest in recent years and many researches are exploring the FMT's potential role for treating other gastrointestinal disease such as IBD. A FMT registry is required to explore the relationship between disease prognosis and intestinal microbiota.

DETAILED DESCRIPTION:
The human intestinal microbiota is composed of complex community of 10*13 to 10*14 commensal microorganisms[1]. Human intestine provides a nutrient-rich habitat for intestinal microorganism which allows a diverse ecosystem to enhance their host's immune system and facilitate digestive activities. Numerous researches are investigating the role of gut microbiota in human homeostasis, which may be related to the pathogenesis of gastrointestinal disease and autoimmune disorder. A research using gene-sequencing technique showed an abnormal microbiota composition such as specific group of Escherichia coli and decreased diversity of intestinal microbiota in individuals with Inflammatory Bowel Disease (IBD) [2-4]. These microbiotas may stimulate the production of cytokine and chemokines that leads to the mucosal inflammatory activity[5]. Gut microbiota may also link with the development of obesity and diabetes by affecting host fat storage and increasing energy harvest from the diet[6-7].

Fecal microbiota transplantation (FMT) is defined as infusion of feces from healthy donors to affected subjects. FMT works by altering the patient's microbiome and it is now recommended as an effective therapy for Clostridium difficile infection (CDI) not responding to standard therapies8. It has attracted great interest in recent years and many researches are exploring the FMT's potential role for treating other gastrointestinal disease such as IBD. A recent clinical study evaluated the efficacy of FMT in active Ulcerative Colitis. It showed one-forth cases of the FMT group were in UC remission and an increase in diversity of microbiota composition. However, these results were dependent on the donor[9].

There will be increasing use of FMT in clinical practice, as well as more studies investigating the effectiveness of FMT on other diseases in the future. However, as an emerging procedure, there is currently no registry system to track patient safety information of FMT. It is also equally important to promote scientific investigation around gut microbiome. Therefore, the investigators aim to establish a FMT registry platform to collect clinical data and specimen from FMT recipients and donors. This registry is initiated Hong Kong, and will be expanded to other part of Asia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Written informed consent obtained
* Subject who has received or planning to receive FMT or other gut-related microbiota products in routine clinical practice or research (FMT recipents)
* Subject who has donated stool or planning to donate stool for FMT or production of other gut-related microbiota products in routine clinical practice or research. Subjects who failed screening will also be recruited. (FMT donors)

Exclusion Criteria:

* Age ≤18

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: FMT Recipients Subject who has received or planning to receive FMT or other gut-related microbiota products in routine clinical practice or research
  FMT Donors Subject who has donated stool or planning to donate stool for FMT or production of other gut-related microbiota products in routine clinical practice or research.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-07-02 (Actual); Primary Completion 2046-05 (Estimated); Study Completion 2046-11 (Estimated)

PRIMARY OUTCOMES:
Set up a FMT registry | 10 years
  Set up a registry of FMT to collect data such as demographics, past medical history, surgery, severity of disease indicated for FMT cases

SECONDARY OUTCOMES:
Patient outcome of FMT | 10 years
  Compare the severity of disease, any adverse event related to FMT and hospitalization between baseline and FMT. Survey
Factors associated with successful FMT | 10 years
  Study samples will collected to characterize which microbiota favors FMT by performing metagenomics of gut microbiome in stool samples
Characterize FMT stool donors and other gut-related microbiota products | 10 years
  Collect study samples to characterize which microbiota favors FMT by metagenomics
FMT in Asia | 10 years
  Gather information such as the severity of disease, any adverse event related to FMT and hospitalization from other study sites in Asia. Survey
Promoting scientific investigation in FMT | 10 years
  Collect study samples to characterize which microbiota favors FMT by metagenomics
Future research studies | 10 years
  Number of patients who may be eligible for participation in future research studies by collecting their information demographics, past medical history, surgery, severity of disease
Developing Biobank of FMT | 10 years
  Collect and store of study samples from recipients and donors to characterize which microbiota favors FMT by metagenomics

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Yau YK, Lau LHS, Lui RNS, Wong SH, Guo CL, Mak JWY, Ching JYL, Ip M, Kamm MA, Rubin DT, Chan PKS, Chan FKL, Ng SC. Long-Term Safety Outcomes of Fecal Microbiota Transplantation: Real-World Data Over 8 Years From the Hong Kong FMT Registry. Clin Gastroenterol Hepatol. 2024 Mar;22(3):611-620.e12. doi: 10.1016/j.cgh.2023.09.001. Epub 2023 Sep 19. PMID 37734581